CLINICAL TRIAL: NCT04843995
Title: The Effect of Mid-urethral Sling on the Urethral Dynamic Shape and Motion
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Other Study IDs: EH21-027
Record Dates: First submitted 2021-04-07; First posted 2021-04-14 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Suburethral Slings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Mid-urethral sling — Treatment of stress urinary incontinence with retropubic mid-urethral sling

SUMMARY:
The purpose of this prospective cohort study is to investigate the effect of sling on urethral dynamic shape and motion using static and dynamic pelvic floor ultrasound and additionally compare the findings among women with successful vs failed surgical outcome.

DETAILED DESCRIPTION:
This study is designed as a prospective cohort study. Our hypothesis is that mid-urethral sling provides backstop for excessive "swing motion" of distal urethra and helps with urethral compression along its luminal axis.

Aim 1: Investigate the effect of mid-urethral sling on the urethral shape at rest and maximum Valsalva, in other words dynamic urethral shape.

Aim 2: Compare the effect of mid-urethral sling on urethral dynamic shape in women with successful surgical outcome (absence of stress urinary incontinence at 3 and 12 months after the surgery) and women with surgical failure (presence of stress urinary incontinence at 3 and 12 months after the surgery).

ELIGIBILITY:
Inclusion Criteria:

* stress urinary incontinence interested in treatment with mid-urethral sling
* able to consent in english and come to post-operative and research visits

Exclusion Criteria:

* contraindication to mid-urethral sling
* detrusor overactivity > 40cm H2O
* post-void residual > 150mL
* Maximum urethral closure pressure < 40 cm H2O

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women over 18 years old with stress urinary incontinence interested in treatment with midurethral sling
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2012-06-11 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Urethral Shape at 3 months | 3 months
  Urethral shape measured by ultrasound
Urethral Motion at 3 months | 3 months
  Urethral motion measured by ultrasound
Urethral Shape at 12 months | 12 months
  Urethral shape measured by ultrasound
Urethral Motion at 12 months | 12 months
  Urethral motion measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Joel D Winer, MD, Principal Investigator — Endeavor Health; Ghazaleh Rostami Nia, MD, Study Chair — Endeavor Health; Henry Chill, MD, Study Director — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Skokie, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richter HE, Albo ME, Zyczynski HM, Kenton K, Norton PA, Sirls LT, Kraus SR, Chai TC, Lemack GE, Dandreo KJ, Varner RE, Menefee S, Ghetti C, Brubaker L, Nygaard I, Khandwala S, Rozanski TA, Johnson H, Schaffer J, Stoddard AM, Holley RL, Nager CW, Moalli P, Mueller E, Arisco AM, Corton M, Tennstedt S, Chang TD, Gormley EA, Litman HJ; Urinary Incontinence Treatment Network. Retropubic versus transobturator midurethral slings for stress incontinence. N Engl J Med. 2010 Jun 3;362(22):2066-76. doi: 10.1056/NEJMoa0912658. Epub 2010 May 17. PMID 20479459
- [Background] Kenton K, Stoddard AM, Zyczynski H, Albo M, Rickey L, Norton P, Wai C, Kraus SR, Sirls LT, Kusek JW, Litman HJ, Chang RP, Richter HE. 5-year longitudinal followup after retropubic and transobturator mid urethral slings. J Urol. 2015 Jan;193(1):203-10. doi: 10.1016/j.juro.2014.08.089. Epub 2014 Aug 23. PMID 25158274
- [Background] Brubaker L, Richter HE, Norton PA, Albo M, Zyczynski HM, Chai TC, Zimmern P, Kraus S, Sirls L, Kusek JW, Stoddard A, Tennstedt S, Gormley EA; Urinary Incontinence Treatment Network. 5-year continence rates, satisfaction and adverse events of burch urethropexy and fascial sling surgery for urinary incontinence. J Urol. 2012 Apr;187(4):1324-30. doi: 10.1016/j.juro.2011.11.087. Epub 2012 Feb 15. PMID 22341290
- [Background] Albo ME, Richter HE, Brubaker L, Norton P, Kraus SR, Zimmern PE, Chai TC, Zyczynski H, Diokno AC, Tennstedt S, Nager C, Lloyd LK, FitzGerald M, Lemack GE, Johnson HW, Leng W, Mallett V, Stoddard AM, Menefee S, Varner RE, Kenton K, Moalli P, Sirls L, Dandreo KJ, Kusek JW, Nyberg LM, Steers W; Urinary Incontinence Treatment Network. Burch colposuspension versus fascial sling to reduce urinary stress incontinence. N Engl J Med. 2007 May 24;356(21):2143-55. doi: 10.1056/NEJMoa070416. Epub 2007 May 21. PMID 17517855
- [Background] Hunskaar S, Lose G, Sykes D, Voss S. The prevalence of urinary incontinence in women in four European countries. BJU Int. 2004 Feb;93(3):324-30. doi: 10.1111/j.1464-410x.2003.04609.x. PMID 14764130
- [Background] Wong V, Shek KL. The mesh debate: Transvaginal anterior anchored mesh should not be abandoned. Aust N Z J Obstet Gynaecol. 2017 Feb;57(1):105-107. doi: 10.1111/ajo.12589. No abstract available. PMID 28251634
- [Background] Ling C, Shek KL, Gillor M, Caudwell-Hall J, Dietz HP. Is location of urethral kinking a confounder of association between urethral closure pressure and stress urinary incontinence? Ultrasound Obstet Gynecol. 2021 Mar;57(3):488-492. doi: 10.1002/uog.22153. PMID 32672377
- [Background] Tamma A, Bjelic-Radisic V, Holbfer S, Trutnovsky G, Tamussino K, Aigmuller T, Ulrich D. Sonographic sling position and cure rate 10-years after TVT- O procedure. PLoS One. 2019 Jan 7;14(1):e0209668. doi: 10.1371/journal.pone.0209668. eCollection 2019. PMID 30615677
- [Background] Milley PS, Nichols DH. The relationship between the pubo-urethral ligaments and the urogenital diaphragm in the human female. Anat Rec. 1971 Jul;170(3):281-3. doi: 10.1002/ar.1091700304. No abstract available. PMID 5104318
- [Background] Stein TA, DeLancey JO. Structure of the perineal membrane in females: gross and microscopic anatomy. Obstet Gynecol. 2008 Mar;111(3):686-93. doi: 10.1097/AOG.0b013e318163a9a5. PMID 18310372